CLINICAL TRIAL: NCT01892722
Title: A 2 Year, Double-blind, Randomized, Multicenter, Active-controlled Core Phase to Evaluate Safety & Efficacy of Daily Fingolimod vs Weekly Interferon β-1a im in Pediatric Patients With Multiple Sclerosis and 5 Year Fingolimod Extension Phase
Brief Title: Safety and Efficacy of Fingolimod in Pediatric Patients With Multiple Sclerosis
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CFTY720D2311; 2011-005677-23 (EudraCT Number)
Record Dates: First submitted 2013-05-08; First posted 2013-07-04 (Estimated); Results first posted 2018-09-19 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-11

CONDITIONS: Multiple Sclerosis
Keywords: pediatric; multiple sclerosis; fingolimod; pre-pubertal; low weight; children; adolescent; MS; core phase; extension phase; younger cohort
MeSH Terms: conditions — Multiple Sclerosis; Thinness | interventions — Interferon beta-1a; Fingolimod Hydrochloride

STUDY DESIGN:
Intervention Model Description: There are 2 arms in the core phase. In the extension phase all participants are receiving open-label.study drug. A third arm has been added to enroll up to 25 new younger patients per HA post approval commitment.
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Fingolimod (Experimental): Fingolimod was administered orally once daily at a dose of either 0.5 mg or 0.25 mg (depending on patient's body weight) with the aim to achieve systemic exposure in range of that in adults at the licensed 0.5 mg dose. Participants in this arm during core continued into extension and received open-label treatment
  Interventions: Drug: Fingolimod; Drug: Placebo capsule
- Interferon beta-1a (Active Comparator): An intramuscular (IM) injection of Interferon beta-1a was administered once weekly during core phase. Participants switched to receive open-label fingolimod in extension phase
  Interventions: Drug: Interferon beta-1a; Drug: Placebo i.m. injection
- Fingolimod-Younger Cohort (Experimental): The 'younger cohort' refers to the new pediatric patients to be recruited in the extension phase who fulfill any single one or a combination of the following criteria: being ≤12 years of age, or weighing ≤40 kg, or being prepubertal (i.e. pubertal status of Tanner stage <2)
  Interventions: Drug: Fingolimod

INTERVENTIONS:
Drug: Interferon beta-1a — Administration once weekly via i.m. injections.
  Arms: Interferon beta-1a
Drug: Fingolimod — Administrated orally once daily:
  0.5 mg capsule for patients over 40 kg or 0.25 mg capsule for patients 40 kg or less.
  Arms: Fingolimod; Fingolimod-Younger Cohort
Drug: Placebo capsule — Matching placebo capsule required for double-dummy masking to blind formulations.
  Arms: Fingolimod
Drug: Placebo i.m. injection — Matching placebo i.m. injection required for double-dummy masking to blind formulations.
  Arms: Interferon beta-1a

SUMMARY:
To evaluate the safety and efficacy of fingolimod vs. interferon beta-1a i.m. in pediatric patients with multiple sclerosis (MS)

DETAILED DESCRIPTION:
The study is divided into a Core Phase, which includes the Double-Blind Treatment Period, and an Extension Phase in which all patients will be treated with fingolimod. The Core Phase is a 24-month, double-blind, randomized, active-controlled, parallel-group multicenter study phase to evaluate the efficacy and safety of fingolimod compared to IFN β-1a in children/adolescent patients aged 10-17 years old with MS. The Extension Phase is a 60-month (5 year) study phase for patients who complete the Core Phase of the study and meet all inclusion/exclusion criteria and for patients who will be recruited in the younger cohort to participate in the Extension Phase. The 'younger cohort' refers to the population of pediatric patients fulfilling any single one or a combination of the following criteria: being ≤12 years of age, or weighing ≤40 kg, or being prepubertal (i.e. pubertal status of Tanner stage <2). The recruitment of the younger cohort (up to 25 patients) was requested as a post- approval health authority commitment

ELIGIBILITY:
Key Inclusion Criteria Core Phase:

* diagnosis of multiple sclerosis
* at least one MS relapse during the previous year or two MS relapses in the previous 2 years or evidence of Gd enhancing lesions on MRI within 6 months EDSS score of 0 to 5.5, inclusive

Key Exclusion Criteria Core Phase:

* patients with progressive MS
* patients with an active, chronic disease of the immune system other than MS
* patients meeting the definition of ADEM
* patients with severe cardiac disease or significant findings on the screening ECG.
* patients with severe renal insufficiency

Key Inclusion Criteria Extension Phase:

Applies to all patients participating in the Core Phase and then entering the Extension Phase. 1. Patients that originally met Core Phase Inclusion criteria and completed the Core phase on or off of study drug.

Applies to patients newly recruited to participate in the Extension Phase.

* All newly recruited patients' that enroll directly into the Extension Phase must fulfill the local country health authority product label approved for pediatric age group for inclusion criteria.
* Central review (including initial MRI report) of the diagnosis of pediatric MS will be required for all newly recruited patients.

Key Exclusion Criteria Extension Phase:

Applies to patients who completed the Core Phase, but prematurely discontinued study drug.

1. Premature discontinuation of the study drug during the Core Phase due to:

   * an adverse event,
   * serious adverse event,
   * laboratory abnormality
   * other conditions leading to permanent study drug discontinuation due to safety reasons
2. Patients with known new events or concomitant medications (washout periods required prior to Visit 15) that would exclude them from the Core Phase exclusion criteria. Serological or other additional tests will not be required.

Applies to patients newly recruited in the younger cohort to participate in the Extension Phase.

1. All newly recruited patients in the younger cohort that enroll directly into the Extension Phase must fulfill the exclusion criteria for the core phase.

Ages: 10 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 240 (Actual)
Dates: Start 2013-07-26 (Actual); Primary Completion 2017-07-14 (Actual); Study Completion 2030-02-18 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (70):
- United States (10):
  - UAB Childrens Hospital Harbor Center Neurology Dept, Birmingham, Alabama
  - Childrens Hospital Los Angeles, Los Angeles, California
  - UCSF, San Francisco, California
  - University of Miami, Miami, Florida
  - AMO Corporation, Tallahassee, Florida
  - Massachusetts General Hospital, Boston, Massachusetts
  - Wayne State University, Detroit, Michigan
  - Robert Wood Johnson Medical School, New Brunswick, New Jersey
  - Childrens Hospital of Philadelphia, Philadelphia, Pennsylvania
  - University of Utah Clinical Trials Office, Salt Lake City, Utah
- Novartis Investigative Site, Parkville, Victoria, Australia
- Novartis Investigative Site, Vienna, Austria
- Brazil (4):
  - Novartis Investigative Site, Belo Horizonte, Minas Gerais
  - Novartis Investigative Site, Rio de Janeiro, Rio de Janeiro
  - Novartis Investigative Site, São Paulo, São Paulo
  - Novartis Investigative Site, Goiânia
- Novartis Investigative Site, Sofia, Bulgaria
- Canada (2):
  - Novartis Investigative Site, Calgary, Alberta
  - Novartis Investigative Site, Ottawa, Ontario
- Novartis Investigative Site, Osijek, Croatia
- Novartis Investigative Site, Tallinn, Estonia
- France (5):
  - Novartis Investigative Site, Bordeaux
  - Novartis Investigative Site, Le Kremlin-Bicêtre
  - Novartis Investigative Site, Marseille
  - Novartis Investigative Site, Montpellier
  - Novartis Investigative Site, Toulouse
- Germany (5):
  - Novartis Investigative Site, Freiburg im Breisgau, Baden-Wurttemberg
  - Novartis Investigative Site, Göttingen, Lower Saxony
  - Novartis Investigative Site, Dresden, Saxony
  - Novartis Investigative Site, Bochum
  - Novartis Investigative Site, Erlangen
- Italy (7):
  - Novartis Investigative Site, Bari, BA
  - Novartis Investigative Site, Montichiari, BS
  - Novartis Investigative Site, Catania, CT
  - Novartis Investigative Site, Milan, MI
  - Novartis Investigative Site, Cefalù, PA
  - Novartis Investigative Site, Roma, RM
  - Novartis Investigative Site, Gallarate, VA
- Novartis Investigative Site, Riga, Latvia
- Novartis Investigative Site, Kaunas, LTU, Lithuania
- Mexico (2):
  - Novartis Investigative Site, Mexico City, D F
  - Novartis Investigative Site, Distrito Federal
- Novartis Investigative Site, Rotterdam, South Holland, Netherlands
- Poland (4):
  - Novartis Investigative Site, Lodz
  - Novartis Investigative Site, Lublin
  - Novartis Investigative Site, Poznan
  - Novartis Investigative Site, Wroclaw
- San Jorge Childrens Hospital, Santurce, Puerto Rico
- Novartis Investigative Site, Bucharest, Romania
- Russia (4):
  - Novartis Investigative Site, Kazan'
  - Novartis Investigative Site, Moscow
  - Novartis Investigative Site, Novosibirsk
  - Novartis Investigative Site, Saint Petersburg
- Novartis Investigative Site, Belgrade, Serbia
- Novartis Investigative Site, Bratislava, Slovakia
- Spain (6):
  - Novartis Investigative Site, Seville, Andalusia
  - Novartis Investigative Site, Vigo, Pontevedra
  - Novartis Investigative Site, Barakaldo, Vizcaya
  - Novartis Investigative Site, Madrid
  - Novartis Investigative Site, Málaga
  - Novartis Investigative Site, Valencia
- Turkey (Türkiye) (5):
  - Novartis Investigative Site, Samsun, Atakum
  - Novartis Investigative Site, Izmir, Balcova
  - Novartis Investigative Site, Istanbul, Fatih
  - Novartis Investigative Site, Ankara, Sihhiye-Altindag
  - Novartis Investigative Site, Ankara, Yenimahalle
- Novartis Investigative Site, Kharkiv, Ukraine
- United Kingdom (3):
  - Novartis Investigative Site, West Midlands, Birmingham
  - Novartis Investigative Site, Edinburgh
  - Novartis Investigative Site, London

IPD SHARING:
Plan to Share IPD: Undecided
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com

REFERENCES:
- [Derived] Deiva K, Huppke P, Banwell B, Chitnis T, Gartner J, Krupp L, Waubant E, Stites T, Pearce GL, Merschhemke M. Consistent control of disease activity with fingolimod versus IFN beta-1a in paediatric-onset multiple sclerosis: further insights from PARADIGMS. J Neurol Neurosurg Psychiatry. 2020 Jan;91(1):58-66. doi: 10.1136/jnnp-2019-321124. Epub 2019 Aug 29. PMID 31467033
- [Derived] Chitnis T, Arnold DL, Banwell B, Bruck W, Ghezzi A, Giovannoni G, Greenberg B, Krupp L, Rostasy K, Tardieu M, Waubant E, Wolinsky JS, Bar-Or A, Stites T, Chen Y, Putzki N, Merschhemke M, Gartner J; PARADIGMS Study Group. Trial of Fingolimod versus Interferon Beta-1a in Pediatric Multiple Sclerosis. N Engl J Med. 2018 Sep 13;379(11):1017-1027. doi: 10.1056/NEJMoa1800149. PMID 30207920
- See also: Recruitment website — https://www.nationalmssociety.org/Research/Participate-in-Research-Studies/Participate-in-Clinical-Trials

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: This study is divided into a core phase and extension phase. In the core phase, patients were randomized to Fingolimod or Interferon beta-1a in a 1:1 ratio. The core phase disposition is reported for interim results disclosure. Upon completion of the extension phase, the extension disposition will be reported.
Groups:
- Fingolimod: Fingolimod was administered orally once daily at a dose of either 0.5 mg or 0.25 mg (depending on patient's body weight) with the aim to achieve systemic exposure in range of that in adults at the licensed 0.5 mg dose.
- Interferon Beta-1a: An intramuscular (IM) injection of Interferon beta-1a was administered once weekly.
Period: Overall Study
Arm/Group | Fingolimod | Interferon Beta-1a
Started | 107 | 108
Full Analysis Set | 107 | 107
Completed | 100 | 88
Not Completed | 7 | 20
Not completed — Protocol deviation | 0 | 1
Not completed — Administrative problems | 0 | 1
Not completed — Patient/guardian decision | 0 | 2
Not completed — Physician Decision | 1 | 2
Not completed — Adverse Event | 3 | 2
Not completed — Lack of Efficacy | 0 | 7
Not completed — Withdrawal by Subject | 3 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Fingolimod | Interferon Beta-1a | Total
Number analyzed (Participants) | 107 | 108 | 215
Age, Continuous [Mean (Standard Deviation); unit: Years] | 15.2 (2.0) | 15.4 (1.60) | 15.3 (1.81)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 70 | 64 | 134
  Male | 37 | 44 | 81
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 3 | 2 | 5
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 4 | 5
  White | 100 | 97 | 197
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 2 | 5 | 7

OUTCOME MEASURES:

1. Primary Outcome: Frequency of Relapses in Patients Treated for up to 24 Months
Description: Frequency of relapses assessed by the annualized relapse rate (ARR). The ARR is defined as the average number of confirmed relapses per year (total number of confirmed relapses divided by the total days in the study multiplied by 365.25).
Time Frame: 24 months
Population: Full analysis set (FAS): The FAS was comprised of all randomized patients with assigned treatments who received at least one dose of study medication.
Measure: Mean (95% Confidence Interval); unit: Confirmed relapse per year
Arm/Group | Fingolimod | Interferon Beta-1a
Number analyzed (Participants) | 107 | 107
Confirmed relapse per year | 0.122 [0.078 to 0.192] | 0.675 [0.515 to 0.885]
Statistical Analysis 1: Comparison: Fingolimod vs Interferon Beta-1a; Test type: Superiority; p < 0.001, Negative binomial regression model

2. Secondary Outcome: New/Newly Enlarged T2 Lesions
Description: Annualized rate of the number of new/newly enlarged T2 lesions up to Month 24
Time Frame: 24 months
Reporting Status: Not Posted, anticipated posting 2030-08

3. Secondary Outcome: Time to First Relapse
Description: Time to first relapse was determined.
Time Frame: 24 months
Reporting Status: Not Posted, anticipated posting 2030-08

4. Secondary Outcome: Proportion of Patients Relapse-free
Description: Proportion of patients relapse-free was determined
Time Frame: 24 months
Reporting Status: Not Posted, anticipated posting 2030-08

5. Secondary Outcome: T1 Gd- Enhancing Lesions
Description: Number of T1 Gd-enhancing lesions per scan up to Month 24
Time Frame: 24 months
Reporting Status: Not Posted, anticipated posting 2030-08

6. Secondary Outcome: Pharmacokinetics (Cavg) of Fingolimod-P
Description: Cavg (average drug concentration over the dose interval) will be evaluated.
Time Frame: 24 months
Reporting Status: Not Posted, anticipated posting 2030-08

7. Secondary Outcome: Pharmacokinetic/Pharmacodynamic Relationship for Fingolimod-P to Lymphocyte Levels
Description: Population PK/PD modeling approaches were used to relate the individual fingolimod-P concentrations to lymphocyte counts.
Time Frame: 24 months
Reporting Status: Not Posted, anticipated posting 2030-08

ADVERSE EVENTS:
Time Frame: Time Frame Adverse Events (AEs) are collected from First Patient First Visit (FPFV) until Last Patient Last Visit (LPLV) for the primary endpoint. All AEs reported in this record are from date of First Patient First Treatment until Last Patient Last Visit for the primary endpoint, up to approximately 4 years. The trial is ongoing.
Arm/Group | Fingolimod | Interferon Beta-1a
All-Cause Mortality (participants affected / at risk) | 0/107 | 0/107
Serious Adverse Events (participants affected / at risk) | 19/107 | 10/107
Other Adverse Events (participants affected / at risk) | 82/107 | 94/107
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Fingolimod (N=107) | Interferon Beta-1a (N=107)
Agranulocytosis (Blood and lymphatic system disorders) | 1 | 0
Leukopenia (Blood and lymphatic system disorders) | 2 | 0
Atrioventricular block second degree (Cardiac disorders) | 1 | 0
Supraventricular tachycardia (Cardiac disorders) | 0 | 1
Autoimmune uveitis (Eye disorders) | 1 | 0
Uveitis (Eye disorders) | 0 | 1
Dyspepsia (Gastrointestinal disorders) | 1 | 0
Gastrointestinal necrosis (Gastrointestinal disorders) | 1 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 1
Rectal tenesmus (Gastrointestinal disorders) | 1 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 1 | 0
Fatigue (General disorders) | 0 | 1
Pyrexia (General disorders) | 0 | 1
Abscess oral (Infections and infestations) | 1 | 0
Appendicitis (Infections and infestations) | 1 | 0
Cellulitis (Infections and infestations) | 1 | 0
Gastritis viral (Infections and infestations) | 0 | 1
Gastrointestinal infection (Infections and infestations) | 1 | 0
Paronychia (Infections and infestations) | 0 | 1
Viral infection (Infections and infestations) | 1 | 0
Viral pharyngitis (Infections and infestations) | 1 | 0
Head injury (Injury, poisoning and procedural complications) | 1 | 0
Humerus fracture (Injury, poisoning and procedural complications) | 1 | 0
Alanine aminotransferase increased (Investigations) | 1 | 0
Body temperature increased (Investigations) | 0 | 1
Gamma-glutamyltransferase increased (Investigations) | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 0
Dizziness (Nervous system disorders) | 0 | 1
Epilepsy (Nervous system disorders) | 1 | 0
Generalised tonic-clonic seizure (Nervous system disorders) | 1 | 0
Headache (Nervous system disorders) | 0 | 1
Migraine (Nervous system disorders) | 1 | 0
Migraine without aura (Nervous system disorders) | 1 | 0
Multiple sclerosis plaque (Nervous system disorders) | 1 | 0
Multiple sclerosis relapse (Nervous system disorders) | 1 | 3
Optic neuritis (Nervous system disorders) | 0 | 1
Seizure (Nervous system disorders) | 2 | 0
Sensory loss (Nervous system disorders) | 0 | 1
Bladder spasm (Renal and urinary disorders) | 1 | 0
Dysuria (Renal and urinary disorders) | 1 | 0
Hypersensitivity vasculitis (Skin and subcutaneous tissue disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Fingolimod (N=107) | Interferon Beta-1a (N=107)
Leukopenia (Blood and lymphatic system disorders) | 14 | 3
Abdominal pain (Gastrointestinal disorders) | 9 | 9
Diarrhoea (Gastrointestinal disorders) | 8 | 10
Nausea (Gastrointestinal disorders) | 9 | 5
Toothache (Gastrointestinal disorders) | 6 | 2
Vomiting (Gastrointestinal disorders) | 8 | 7
Chills (General disorders) | 1 | 11
Fatigue (General disorders) | 10 | 6
Influenza like illness (General disorders) | 5 | 40
Pyrexia (General disorders) | 8 | 21
Influenza (Infections and infestations) | 12 | 4
Nasopharyngitis (Infections and infestations) | 8 | 5
Rhinitis (Infections and infestations) | 10 | 9
Upper respiratory tract infection (Infections and infestations) | 17 | 5
Viral upper respiratory tract infection (Infections and infestations) | 23 | 26
Glomerular filtration rate decreased (Investigations) | 1 | 6
White blood cell count decreased (Investigations) | 6 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 6 | 6
Headache (Nervous system disorders) | 34 | 31
Anxiety (Psychiatric disorders) | 7 | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 10 | 12
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 9 | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial or disclosure of trial results in their entirety.

DOCUMENTS (2):
  • Study Protocol (2016-11-16): https://cdn.clinicaltrials.gov/large-docs/22/NCT01892722/Prot_001.pdf
  • Statistical Analysis Plan (2017-08-04): https://cdn.clinicaltrials.gov/large-docs/22/NCT01892722/SAP_000.pdf